CLINICAL TRIAL: NCT07134049
Title: Investigation of the Effects of Sensory Integration Therapy on Sensory, Motor, and Cognitive Development in Children With Congenital Brachial Plexus Injury
Brief Title: Sensory Integration Therapy in Children With Congenital Brachial Plexus Injury: Developmental Outcomes
Acronym: SI-BPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Cimilli, MSc, Principal Investigator, Occupational Therapist (MSc), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-68552689-000-00004173157; Hacettepe University (Other: Hacettepe University)
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Obstetric Brachial Plexus Injury
Keywords: sensory integration; Cognitive development; Motor development; obstetric brachial plexus palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in this group receive individualized sensory integration therapy sessions once a week for 8 weeks, in addition to their routine physiotherapy program. Each session lasts approximately 45 minutes and is based on the core principles of sensory integration therapy. The intervention includes activities involving tactile, vestibular, proprioceptive, auditory, and visual stimuli, tailored to each child's sensory processing needs. Therapy is provided in a sensory-enriched and safe environment, and aims to promote adaptive responses, motor planning, self-regulation, and functional skills. Sessions are play-based and structured to support engagement and motivation.
  Interventions: Other: sensory integration therapy
- control group (No Intervention): Participants in this group will not receive any sensory integration therapy during the 8-week study period. Instead, they will continue with their existing routine physiotherapy program, which may include general motor exercises, range of motion activities, and other standard therapeutic practices. No additional sensory-based interventions will be introduced. This group serves as a comparator to assess the effects of sensory integration therapy provided to the experimental group

INTERVENTIONS:
Other: sensory integration therapy — Sensory Integration Therapy (SIT) is a client-centered rehabilitation approach aimed at improving adaptive and functional responses to sensory stimuli in changing environments. It is based on structured, individualized activities conducted in enriched sensory environments. These environments are designed to be engaging and motivating for children through the use of interactive and playful tasks that match their sensory processing profiles.
  Sensory integration plays a key role in motor planning, postural control, attention, and emotional regulation. Deficits in sensory integration-particularly in vestibular, tactile, and proprioceptive systems-may result in poor muscle tone, difficulty with balance and coordination, and impaired motor planning. These issues can negatively impact the development of gross motor, fine motor, language, and academic skills. For this reason, sensory-based interventions that support neural organization and promote adaptive responses are commonly recommended i
  Arms: intervention group

SUMMARY:
The purpose of this study is to investigate the effectiveness of sensory integration therapy in reducing sensory, motor, and cognitive developmental impairments following Congenital Brachial Plexus Injury (CBPI), and to support the overall developmental processes of affected children.

DETAILED DESCRIPTION:
Detailed Description:

Congenital Brachial Plexus Injury (CBPI) is a peripheral nerve injury occurring during childbirth that can lead to varying degrees of sensory, motor, and functional impairments. These impairments may adversely affect not only motor skills but also sensory processing and cognitive development, particularly in early childhood when neurodevelopment is highly plastic. Sensory integration therapy is a child-centered, play-based intervention designed to improve the brain's ability to process and integrate sensory information from the tactile, vestibular, proprioceptive, visual, and auditory systems. By providing enriched and graded sensory experiences, this therapeutic approach aims to promote adaptive responses, improve motor planning, enhance self-regulation, and support overall developmental progress.

The purpose of this study is to evaluate the effectiveness of sensory integration therapy in reducing sensory, motor, and cognitive developmental impairments in children with CBPI aged 7 to 35 months. Participants in the intervention group will receive individualized sensory integration therapy sessions once a week for 8 weeks, in addition to their routine physiotherapy programs. Developmental outcomes will be assessed using standardized assessment tools before and after the intervention. The findings of this study are expected to contribute to evidence-based rehabilitation approaches for children with CBPI and to inform early intervention strategies aimed at optimizing sensory, motor, and cognitive development.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of obstetric brachial plexus injury (OBPI) Age between 7 and 35 months No additional diagnosed neurological, psychiatric, and/or muscular disorders No diagnosed mental retardation or cognitive disorder that would prevent participation in assessments Written informed consent from parents or legal guardians

Exclusion Criteria:

Severe visual or hearing impairment preventing participation in assessments Participation in another experimental rehabilitation program within the last 3 months

Ages: 7 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) | The assessment will be conducted at the beginning of the treatment and repeated at the end of the 8-week treatment period.
  The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) is a standardized assessment tool designed to evaluate the developmental functioning of infants and toddlers aged 1 to 42 months. It measures five key domains: Cognitive, Language (Receptive and Expressive), Motor (Fine and Gross), Social-Emotional, and Adaptive Behavior.
  The Bayley-III is widely used in clinical and research settings to identify developmental delays and to monitor developmental progress over time

SECONDARY OUTCOMES:
Dunn Infant/Toddler Sensory Profile (7-35 months) | The assessment will be conducted at the beginning of the treatment and repeated at the end of the 8-week treatment period.
  The Dunn Infant/Toddler Sensory Profile is a standardized caregiver questionnaire designed to assess sensory processing patterns in infants and toddlers aged 7 to 35 months. Developed by Winnie Dunn, the tool evaluates how young children respond to sensory experiences in their daily environments, based on caregiver observations.
Active Movement Scale (AMS) | The assessment will be conducted at the beginning of the treatment and repeated at the end of the 8-week treatment period
  The Active Movement Scale (AMS) is a standardized clinical assessment tool used to evaluate voluntary motor function in infants and young children, particularly those with brachial plexus birth injury (BPBI) or other upper limb neuromuscular impairments.
  The AMS is designed for children from birth up to 1 year of age and beyond, depending on developmental stage. It assesses active range of motion (AROM) in the upper extremities, both against gravity and with gravity eliminated.
Modified Mallet Grading System (MMGS) | he assessment will be conducted at the beginning of the treatment and repeated at the end of the 8-week treatment period.
  The Modified Mallet Grading System (MMGS) is a clinical assessment tool used to evaluate shoulder function in patients with brachial plexus birth palsy (BPBP). It measures the functional range and quality of specific shoulder movements through observation of task-based activities.
  The MMGS is widely used due to its simplicity, reliability, and ability to track surgical and therapeutic outcomes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Öksüz, PhD, Professor,, Principal Investigator — Hacettepe University Faculty of Health Sciences, Department of Occupational Therapy
Locations (1):
- Hacettepe Univeristy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared